CLINICAL TRIAL: NCT00299819
Title: A Phase I, Randomized, Double-Blind, Placebo Controlled, Dose-Escalation Study to Evaluate Safety and Tolerability of a Single IV Dose of MEDI-545, a Fully Human Monoclonal Antibody Directed Against Interferon Alpha Subtypes, in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Safety and Tolerability of MEDI-545 in Patients Who Have Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Greg Dennis, M.D., MedImmune Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP126; NCT00394719 (obsolete NCT alias)
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Lupus
Keywords: Lupus
MeSH Terms: interventions — sifalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Active Comparator): MEDI-545
  Interventions: Biological: MEDI 545
- 2 (Active Comparator): MEDI-545
  Interventions: Biological: MEDI-545
- 3 (Active Comparator): MEDI-545
  Interventions: Biological: MEDI-545
- 4 (Active Comparator): MEDI-545
  Interventions: Biological: MEDI-545
- 5 (Active Comparator): MEDI-545
  Interventions: Biological: MEDI-545

INTERVENTIONS:
Biological: MEDI-545 — 0.3 mg/kg IV (n=6) at Study Day 0
  Arms: 2
Biological: MEDI 545 — 0.3 mg/kg IV (n=6) at Study Day 0
  Arms: 1
Biological: MEDI-545 — 0.3 mg/kg IV (n=6) at Study Day 0
  Arms: 3
Biological: MEDI-545 — 0.3 mg/kg IV (n=6) at Study Day 0
  Arms: 4
Biological: MEDI-545 — 0.3 mg/kg IV (n=6) at Study Day 0
  Arms: 5

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of intravenously administered MEDI-545 compared with placebo, over a dose escalation range of 0.3-30 mg/kg, in adult patients with SLE and who are receiving 20 mg/day or less of prednisone orally or an equivalent dose of another oral corticosteroid.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of intravenously administered MEDI-545 compared with placebo, over a dose escalation range of 0.3-30 mg/kg, in adult patients who have SLE and who are receiving 20 mg/day or less of prednisone orally or an equivalent dose of another oral corticosteroid.

The secondary objective of this study is to describe the pharmacokinetics and potential immunogenicity of MEDI-545.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria:
* Adult males and females ≥ 18 years at the time of the first dose of study drug.
* Written informed consent obtained from the patient/patient's legal guardian
* Diagnosis of SLE: Patients must have previously met ≥ 4 of the 11 revised ACR criteria
* Current background treatments may include the following medications prior to randomization: acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), and antimalarials, such as hydroxychloroquine ≤ 600 mg/day, and prednisone ≤ 20 mg daily (or an equivalent dose of another oral corticosteroid) for at least 28 days
* Sexually active females, unless surgically sterile or at least two years post-menopausal, must use an effective method of avoiding pregnancy (including oral, injectable, transdermal, or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 28 days before the first dose of study drug, and must agree to continue using such precautions through the study period of 84 days. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active males, unless surgically sterile, must likewise use an effective method of birth control (condom or abstinence) and must agree to continue using such precautions through Study Day 84.
* Ability to complete follow-up period of 84 days as required by the protocol.

Exclusion Criteria:

* Weight ≥ 120 kg
* Use of cyclophosphamide, azathioprine, methotrexate, mycophenolate mofetil or cyclosporine within 28 days before study entry
* Use of doses of corticosteroids higher than the equivalent of prednisone 20 mg/day (or an equivalent dose of another corticosteroid) within 28 days before study entry
* In the opinion of the investigator, a likelihood of requiring initiation of immunosuppressant therapy (e.g., prednisone >20 mg daily (or an equivalent dose of another oral corticosteroid), azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, or dapsone) within the 28 days after study entry. Antimalarial dosing must be held constant during the study, but analgesics and NSAIDs may be varied.
* Current treatment with coumadin
* Treatment with immunoglobulin or blood products within 28 days before entry into the study
* Treatment with any investigational drug therapy within 28 days before entry into the study; in the case of cell-depleting therapies, such as B or T cell depletion, cell counts that remain below acceptable or baseline levels (use of licensed agents for indications not listed in the package insert is permitted)
* History of primary immunodeficiency
* History of allergic reactions likely to be exacerbated by any component of the study drug
* Previous medical history, or evidence, of an intercurrent illness, other than SLE, that may compromise the safety of the patient in the study
* Clinically significant cardiac disease, including: unstable angina; myocardial infarction within 6 months; congestive heart failure; arrhythmia requiring active therapy, with the exception of clinically insignificant extra systoles, or minor conduction abnormalities; and history of clinically significant abnormality on electrocardiogram
* Evidence of significant active infection, or vaccination with live attenuated viruses, currently or in the 2 weeks before randomization
* Evidence of infection with hepatitis B or C virus, or HIV-1 or HIV-2, or active infection with hepatitis A, as determined by results of testing at screening
* A history of severe infection with viruses of the herpes family including Epstein-Barr virus requiring hospitalization, disseminated herpes, herpes encephalitis, ophthalmic herpes, or cytomegalovirus
* Herpes zoster ≤ 3 months prior to screening
* Current suppressive antiviral therapy for herpes or other viral infections
* Ongoing, chronic infectious disease such as chronic renal infection or chronic chest infection with bronchiectasis or sinusitis
* Pregnancy (females, unless surgically sterile or at least two years post-menopausal must have a negative serum pregnancy test within 14 days before receiving the study drug and a negative urine pregnancy test on Study Day 0 before receiving the study drug)
* Nursing mother
* History of alcohol or drug abuse within the past 2 years
* Presence of end-stage renal disease, or rapidly progressive glomerulonephritis
* Active central nervous system lupus
* History of stroke, or any cerebrovascular disease requiring medication/treatment.
* History of cancer, apart from basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy >1 year prior to enrollment
* At screening (must be within14 days before entry into the study) any of the following:

  * AST > 1.5x upper limit of normal range (ULN)
  * ALT > 1.5x ULN
  * creatinine > 1.5x ULN for patient's age, sex and weight
  * serum K above or below the normal range
  * hemoglobin < 8 g/dL
  * white blood cell count < 1,800/mm3 (Superscript)
  * neutrophils < 1,500/mm3 (Superscript)
  * platelet count < 50,000/mm3 (Superscript)
  * other abnormal laboratory values in the screening panel that in the opinion of the principal investigator are judged to potentially confound analysis of study results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MEDI-545 will be assessed primarily by summarizing adverse events. | Day 84

SECONDARY OUTCOMES:
Evaluation of MEDI-545 pharmacokinetics and possible immunogenicity | Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Barbara White, M.D., Study Director — MedImmune LLC
Locations (21):
- United States (19):
  - Pinnacle Research Group, Anniston, Alabama
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Center for Rhematology, Immunology, and Arthritis, Fort Lauderdale, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Tampa Florida Medical Research Group, Tampa, Florida
  - Florida Medical Clinic, Clinical Research Division, Zephyrhills, Florida
  - Louisiana State University Health Sciences Center-Shreveport, Shreveport, Louisiana
  - Johns Hopkins University, School of Medicine, Baltimore, Maryland
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington Div. of Rhematology, Seattle, Washington
  - Center for Innovative Therapy, UCSD School of Medicine, Milwaukee, Wisconsin
  - Froedtert Hospital, Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Merrill JT, Wallace DJ, Petri M, Kirou KA, Yao Y, White WI, Robbie G, Levin R, Berney SM, Chindalore V, Olsen N, Richman L, Le C, Jallal B, White B; Lupus Interferon Skin Activity (LISA) Study Investigators. Safety profile and clinical activity of sifalimumab, a fully human anti-interferon alpha monoclonal antibody, in systemic lupus erythematosus: a phase I, multicentre, double-blind randomised study. Ann Rheum Dis. 2011 Nov;70(11):1905-13. doi: 10.1136/ard.2010.144485. Epub 2011 Jul 27. PMID 21798883
- [Derived] Yao Y, Richman L, Higgs BW, Morehouse CA, de los Reyes M, Brohawn P, Zhang J, White B, Coyle AJ, Kiener PA, Jallal B. Neutralization of interferon-alpha/beta-inducible genes and downstream effect in a phase I trial of an anti-interferon-alpha monoclonal antibody in systemic lupus erythematosus. Arthritis Rheum. 2009 Jun;60(6):1785-96. doi: 10.1002/art.24557. PMID 19479852